CLINICAL TRIAL: NCT05557786
Title: The Treatment of Transcranial Alternating Current Stimulation（tACS）on Patients With Cerebellar Ataxia: A Randomized, Triple-blind, Parallel-controlled Study
Brief Title: Treatment of Transcranial Alternating Current Stimulation（tACS）on Cerebellar Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ning Wang, MD., PhD., Director, First Affiliated Hospital of Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRCTA, ECFAH of FMU[2022]399
Record Dates: First submitted 2022-09-24; First posted 2022-09-28 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Spinocerebellar Ataxia Type 3; Multiple System Atrophy-cerebellar Type
Keywords: SCA3; MSA-C; tACS; Brain oscillations; effectiveness
MeSH Terms: conditions — Machado-Joseph Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real cerebellar tACS for Cerebellar Ataxia (Part Ⅰ: SCA3, Part Ⅱ: MSA-C) (Active Comparator): Real cerebellar tACS, 70Hz, 2mA (peak to peak), 40min/day (10s ramp up and 10s ramp down), (10 sessions, 5 days/week for 2 weeks)
  Interventions: Device: Transcranial Alternating Current Stimulation
- Sham cerebellar tACS for Cerebellar Ataxia (Part Ⅰ: SCA3, Part Ⅱ: MSA-C) (Sham Comparator): Device: Sham cerebellar tACS, 10Hz, 2mA (peak to peak) for 40s, and then no current 40min/day (10s ramp up and 10s ramp down), (10 sessions, 5 days/week for 2 weeks)
  Interventions: Device: Transcranial Alternating Current Stimulation

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation — Cerebellar Transcranial Alternating Current Stimulation（tACS）

SUMMARY:
This is a longitudinal, triple-blind, randomized-controlled, prospective interventional study assessing patients with cerebellar ataxia, including spinocerebellar ataxia type 3 (SCA3) and multiple system atrophy-cerebellar type (MSA-C), to examine the efficacy, safety, and tolerability of transcranial alternating current stimulation (tACS) for up to 3 months.

DETAILED DESCRIPTION:
Transcranial alternating current stimulation (tACS) is a relatively recent method that noninvasively modulates brain oscillations, and can effectively stimulate deep brain regions, affect brain rhythm, increase neural plasticity, change neurotransmitter levels, and improve brain function. It is a comfortable, safe, effective, non-invasive, and easy-to-operate method, which means it has development potential in relevant medical fields. It has been approved by the FDA for clinically treating neuropsychiatric diseases.

This is a prospective, longitudinal, triple-blind, randomized-controlled, interventional study designed to evaluate the efficacy, safety, and tolerability of tACS in patients of SCA3 and MSA-C in China. Based on typical guidelines, we will use the tACS paradigm (bilateral mandible as a place for active electrode stimulation electrode, and the inion for the return electrode). This study has two parts. The patients studied in the Part Ⅰ are SCA3. The patients studied in the Part Ⅱ are MSA-C. Every part of study, subjects will be randomized into two groups, one receiving a 10-day (5 days/week for 2 weeks) treatment with real cerebellar tACS (CB-tACS) and the other receiving a sham stimulation. The patient's motor function, cognitive function, sleep, mental state, plantar pressure, and magnetic resonance imaging will be assessed before and after the intervention.

There will be a total of 4 visits. All patients receiving tACS will be visited face to face at baseline, day 1, day 30, and day 90 after the treatment begins.

ELIGIBILITY:
Inclusion Criteria:

* for SCA3

  * Patients with detectable clinical signs and confirmed genetic diagnosis with SCA3
  * SCA3 patients aged 18 - 80 years
  * Patients or their family members have informed consent to the study and signed relevant documents
  * The pre-study ataxia Assessment Score (SARA) ranged from 3 to 30
* for MSA-C

  * Aged 30-80 years
  * Diagnosed as clinically determined (Established)MSA-C or clinically Probable MSA-C according to the latest MSA diagnostic criteria
  * No more than 8 years after diagnosis of MSA-C
  * Able to walk independently or with assistance
  * Have a life expectancy of at least 3 years
  * Women of childbearing age with MSA need to use contraceptive measures

Exclusion Criteria:

1. Patients who have concomitant epilepsy.
2. Patients with a serious cognitive disorder, behavioral disorder, or mental illness
3. Patients with a history of seizures, stroke, encephalitis, or other degenerative neurological diseases
4. Patients with a serious medical disease

   * Patients who concomitantly suffer from severe renal impairment, convulsions, stomach ulcers, or moderate or more severe liver disease
   * Patients with uncontrolled high blood pressure or diabetes
5. History of head injury or neurosurgical interventions.
6. History of any metal in the head (outside the mouth).
7. Known history of any metallic particles in the eye, implanted cardiac pacemaker, implanted neurostimulators, surgical clips (above the shoulder line), or any medical pumps.
8. Patients who have taken other investigational products within 4 weeks before being enrolled in this clinical trial, or patients who are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2022-08-07 (Actual); Primary Completion 2024-03-09 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
For Part Ⅰ (SCA3) -1 | Baseline - 2 weeks
  To compare the proportion of patients with SARA improvement (decrease) of at least 1.5 from baseline after 2 weeks, assessing changes in the Assessment and Rating of Ataxia (SARA) Score.
For Part Ⅱ (MSA-C) -1 | Baseline - 2 weeks
  Changes of Clinical Evaluation for (Unified Multiple System Atrophy Rating Scale) UMSARS improvement (decrease) from baseline to 2 weeks.
  UMSARS I: This is an assessment of daily life activities via 12 items scale used to assess language, writing, autonomy, walking, and the presence of possible urinary, sexual, or intestinal disorders. (0=no disorder, 48=severe) UMSARS II: Motor examination based on 14 items that evaluate particular facial expression, oculomotricity, oral expression, tremors, or walking. 0= no disorder, 56=severe disorders.
  UMSARS III: Blood pressure and heart rate measurements in lying and standing positions for 10 min every minute.
  UMSARS IV: Assessment of the disability from 1 to 5; 1 = completely independent; 5 = totally dependent.

SECONDARY OUTCOMES:
For Part Ⅰ SCA3 -2 | 1 month - 3 months
  To compare the proportion of patients with SARA improvement (decrease) of at least 1.5 from baseline after 1 month and 3 months, assessing changes in the SARA Score.
For Part Ⅰ SCA3 -3 | Baseline - 2 weeks - 1 month - 3 months
  Changes in the Scale for the SARA improvement (decrease) from baseline to 2 weeks, 1 month and 3 months.
For Part Ⅰ SCA3 -4 | Baseline - 2 weeks - 1 month - 3 months
  Changes in the Scale for the 5 Level EQ-5D (EQ-5D-5L) improvement (decrease) from baseline to 2 weeks, 1 month and 3 months.
  The EQ-5D-5L is a standard measure of health-related quality of life. EQ-5D-5L consists of two components: a health state profile and a visual analog scale (VAS). EQ-5D health state profile comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The 5D-5L systems are converted into a single index utility score between 0 to 1, where a higher score indicates a better health state. The VAS records the participant's health on a 0-100 mm VAS scale, with 0 indicating "the worst health you can imagine" and 100 indicating "the best health you can imagine." Higher scores of EQ-VAS indicate better health.
For Part Ⅱ MSA-C -2 | 1 month - 3 months
  Changes in the Scale for the UMSARS improvement (decrease) from baseline to 1 month and 3 months.
For Part Ⅱ MSA-C -3 | Baseline - 2 weeks - 1 month - 3 months
  Changes in the Scale for the UMSARS II improvement (decrease) from baseline to 2 weeks, 1 month and 3 months.
For Part Ⅱ MSA-C -4 | Baseline - 2 weeks - 1 month - 3 months
  Changes in the Scale for the SARA improvement (decrease) from baseline to 2 weeks, 1 month and 3 months.
For Part Ⅱ MSA-C -5 | Baseline - 2 weeks - 1 month - 3 months
  Changes in the Scale for the Autonomic Scale for Outcomes in Parkinson's Disease (SCOPA-AUT) Score improvement (decrease) from baseline to 2 weeks, 1 month and 3 months.
For Part Ⅱ MSA-C -6 | Baseline - 2 weeks - 1 month - 3 months
  Changes in the Scale for the Multiple System Atrophy Quality of Life (MSA-QoL) Score improvement (decrease) from baseline to 2 weeks, 1 month and 3 months.
  The score of other sub-dimension of the MSA Quality of Life scale. The MSA-QoL questionnaire is composed of three different subscales: motor (14 items), non-motor (12 items), and emotional/social (14 items). The response options for each question range from 0 (no problem) to 4 (extreme problem), with higher total scores reflecting more impaired quality of life. The MSA-QoL also includes a visual analog scale (VAS) of how satisfied patients feel (range 0-100, with lower scores indicating a lower quality of life).

OTHER OUTCOMES:
For SCA3 and MSA-C | Baseline-2 weeks - 1 month - 3 months
  Changes in the temporospatial parameters of gait from baseline to 2 weeks, 1 month and 3 months.
  Gait parameters measured by Multimodal Gait Analysis System. The kinetic and kinematic data of gait will be collected in the gait analysis corridor using two sets of smart insole systems and two sets of gyroscope sensor systems.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, The First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Chen X, Liu X, Lin W, Zhang L, Cheng X, Huang Z, Zhang W, Zeng H, Lian Y, Zhang Y, Li M, Chen N, Huang S, Wang Z, Wang X, Liu Z, Yuan R, Chen X, Ye Z, Cheng B, Zhang Y, Chen Q, Wang D, Ni J, Wang N, Fu Y, Gan S; OSCCAR Investigators. Transcranial alternating current stimulation for treating spinocerebellar ataxia type 3: A randomized controlled trial. Cell Rep Med. 2025 Jun 17;6(6):102162. doi: 10.1016/j.xcrm.2025.102162. PMID 40532663
- [Derived] Liu X, Lin W, Zhang L, Zhang WL, Cheng XP, Lian YH, Li MC, Wang SZ, Chen XY, Gan SR. Effects of cerebellar transcranial alternating current stimulation in cerebellar ataxia: study protocol for a randomised controlled trial. Front Neurosci. 2023 Apr 27;17:1180454. doi: 10.3389/fnins.2023.1180454. eCollection 2023. PMID 37179566

DOCUMENTS (1):
  • Study Protocol (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT05557786/Prot_000.pdf